CLINICAL TRIAL: NCT04730297
Title: Comparative Analgesic Effects of Preoperative Administration of Paracetamol (Acetominophen) 500 mg Plus Codeine 30 mg and Ibuprofen 400 mg on Pain After Third Molar Surgery
Brief Title: Comparative Analgesic Effects of Paracetamol/Codeine and Ibuprofen on Pain After Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Maria Paola Cristalli, Associate Professor DDS, PhD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2704/2013
Record Dates: First submitted 2021-01-13; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: To Control Pain After Third Molar Surgery
Keywords: postsurgical dental pain
MeSH Terms: interventions — Acetaminophen; Codeine; Ibuprofen

STUDY DESIGN:
Intervention Model Description: a single-center, 2-stage, prospective, randomized, triple-blind parallel-group, placebo-controlled, clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paracetamol/codeine Group A (Active Comparator): analgesic group preoperative oral dose of paracetamol 500 mg plus codeine 30 mg
  Interventions: Drug: paracetamol 500 mg plus codeine 30 mg preoperative administration
- Ibuprofen Group B (Active Comparator): analgesic group preoperative oral dose of ibuprofen 400 mg
  Interventions: Drug: ibuprofen 400 mg preoperative administration
- Placebo Group C (Placebo Comparator): Placebo group preoperative placebo
  Interventions: Drug: Placebo oral tablet preoperative administration

INTERVENTIONS:
Drug: paracetamol 500 mg plus codeine 30 mg preoperative administration — each patient 30 minutes before surgery received paracetamol 500 mg plus codeine 30 mg
  Other Names: GROUP A
  Arms: Paracetamol/codeine Group A
Drug: ibuprofen 400 mg preoperative administration — each patient 30 minutes before surgery received ibuprofen 400 mg
  Other Names: GROUP B
  Arms: Ibuprofen Group B
Drug: Placebo oral tablet preoperative administration — each patient 30 minutes before surgery received placebo
  Other Names: GROUP C
  Arms: Placebo Group C

SUMMARY:
To compare analgesic effects of preoperative administration of paracetamol 500 milligram plus codeine 30 milligram in single-tablet and effervescent formulation to ibuprofen 400 milligram, and placebo in the management of moderate to severe postoperative pain after mandibular third molar surgery.

DETAILED DESCRIPTION:
Materials and methods: One hundred twenty healthy outpatients aged 15 to 29 years undergoing surgical removal of one bony impacted mandibular third molar were enrolled in this, single-center, prospective, randomized, triple-blind parallel-group, placebo-controlled, clinical trial. Study participants were randomly assigned to three treatment arms. According to the concealed allocation, each patient 30 minutes before surgery received paracetamol 500 mg plus codeine 30 mg (group A), ibuprofen 400 mg (group B) or placebo (group C). Rescue therapy allowed in the postoperative period was paracetamol 500 mg plus codeine 30 mg in groups A and C and ibuprofen 400 mg in group B. Patients recorded on Numerical Rating Scale-11 (NRS-11) the pain intensity, total number of postoperative-supplement medications and time of the first intake, until 12-hours after surgery and over extra two days

ELIGIBILITY:
Inclusion Criteria:

* healthy status (ASA class I);
* nonsmoker;
* not pregnant or breastfeeding;
* no medication consumption in the past 21 days;
* good oral hygiene;
* bony impaction of one mandibular third molars;
* the presence of the first and second molars;
* compliance to cooperate with the research protocol.

Exclusion Criteria:

* chronic systemic disease;
* medications with potential interaction to paracetamol-codeine or ibuprofen;
* a history of intolerance or hypersensitivity to the study drugs;
* any pre-existing pain and acute inflammatory or infectious conditions; - inability to understand or perform the study procedure.

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) | All study participants were asked to record the pain intensity score at 1:00 pm during the operative day]
  In stage 1, the objective was to misure the efficacy on pain and tolerability of a single dose of paracetamol plus codeine, ibuprofen, or placebo in the operative day. Before surgery, patients were instructed to complete the Numerical Rating Scale-11 (NRS-11), which consisted of an interval scale ranging from 0 ("no pain") to 10 ("maximum pain")
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) | All study participants were asked to record the pain intensity score at 6:00 pm during the operative day]
  In stage 1, the objective was to compare the efficacy on pain and tolerability of a single
  dose of paracetamol plus codeine, ibuprofen, or placebo in the operative day.
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) | All study participants were asked to record the pain intensity score at 11:00 pm during the operative day]
  In stage 1, the objective was to compare the efficacy on pain and tolerability of a single dose of paracetamol plus codeine, ibuprofen, or placebo in the operative day.
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) | All study participants were asked to record the pain intensity score at 8:00 am during the 2th day after surgery]
  In stage 1, the objective was to compare the efficacy on pain and tolerability of a single dose of paracetamol plus codeine, ibuprofen, or placebo
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) | All study participants were asked to record the pain intensity score at 1:00 pm during the 2th day after surgery]
  In stage 1, the objective was to compare the efficacy on pain and tolerability of a single dose of paracetamol plus codeine, ibuprofen, or placebo
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) | All study participants were asked to record the pain intensity score at 6:00 pm during the 2th day after surgery]
  In stage 1, the objective was to compare the efficacy on pain and tolerability of a single dose of paracetamol plus codeine, ibuprofen, or placebo
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) | All study participants were asked to record the pain intensity score at 11:00 pm during the 2th day after surgery]
  In stage 1, the objective was to compare the efficacy on pain and tolerability of a single dose of paracetamol plus codeine, ibuprofen, or placebo in the operative day.
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) | All study participants were asked to record the pain intensity score at 8:00 am during the 3th day after surgery]
  In stage 1, the objective was to compare the efficacy on pain and tolerability of a single dose of paracetamol plus codeine, ibuprofen, or placebo in the operative day.
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) | All study participants were asked to record the pain intensity score at 1:00 pm during the 3th day after surgery]
  In stage 1, the objective was to compare the efficacy on pain and tolerability of a single dose of paracetamol plus codeine, ibuprofen, or placebo in the operative day.
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) | All study participants were asked to record the pain intensity score at 6:00 pm during the 3th day after surgery]
  In stage 1, the objective was to compare the efficacy on pain and tolerability of a single dose of paracetamol plus codeine, ibuprofen, or placebo in the operative day.
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) | All study participants were asked to record the pain intensity score at 11:00 pm during the 3th day after surgery]
  In stage 1, the objective was to compare the efficacy on pain and tolerability of a single dose of paracetamol plus codeine, ibuprofen, or placebo in the operative day.

SECONDARY OUTCOMES:
Number of patients requiring rescue therapy | until 12-hours after surgery and over extra two days
  outcomes involved the number of patients requiring rescue therapy
first postoperative use of analgesics | until 12-hours after surgery
  time of the first intake
total postoperative use of analgesics | until 12-hours after surgery and over extra two days
  total amount of additional medication

OTHER OUTCOMES:
Compare the efficacy of the same drugs | up to 48 hours after stage 1
  Patients recorded on Numerical Rating Scale-11 (NRS-11) the pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Maria Paola Cristalli, DDS, PhD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Maria Paola Cristalli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] La Monaca G, Pranno N, Annibali S, Polimeni A, Pompa G, Vozza I, Cristalli MP. COMPARATIVE ANALGESIC EFFECTS OF SINGLE-DOSE PREOPERATIVE ADMINISTRATION OF PARACETAMOL (ACETAMINOPHEN) 500 mg PLUS CODEINE 30 mg AND IBUPROFEN 400 mg ON PAIN AFTER THIRD MOLAR SURGERY. J Evid Based Dent Pract. 2021 Dec;21(4):101611. doi: 10.1016/j.jebdp.2021.101611. Epub 2021 Jul 10. PMID 34922726